CLINICAL TRIAL: NCT07395895
Title: Effect of Metformin Iontophoresis Combined With Physical Therapy Rehabilitation on Knee Osteoarthritis in Postmenopausal Women: A Randomized Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Effect of Metformin Iontophoresis on Knee Osteoarthritis in Postmenopausal Women
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Eman Said Sawan, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00014233-66
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis in Postmenopausal Women
Keywords: Metformin gel; Iontophoresis; Physical Therapy Rehabilitation; Osteoarthritis; Postmenopausal Women
MeSH Terms: conditions — Osteoarthritis | interventions — Iontophoresis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin Iontophoresis (Active Comparator)
  Interventions: Drug: Metformin gel Iontophoresis
- Iontophoresis Combined with Physical Therapy Rehabilitation (Active Comparator)
  Interventions: Device: Iontophoresis

INTERVENTIONS:
Drug: Metformin gel Iontophoresis — Metformin gel 2% Iontophoresis Combined with Physical Therapy Rehabilitation
  Arms: Metformin Iontophoresis
Device: Iontophoresis — Iontophoresis with neutral gel Combined with Physical Therapy Rehabilitation
  Arms: Iontophoresis Combined with Physical Therapy Rehabilitation

SUMMARY:
This study is designed as a randomized, double-blind, placebo-controlled clinical trial with two parallel groups. All participants will receive a standardized physical therapy rehabilitation program. Participants will be randomly allocated into either a study group receiving metformin iontophoresis or a control group receiving placebo iontophoresis. Both participants and outcome assessors will be blinded to group allocation.

DETAILED DESCRIPTION:
The study population will consist of postmenopausal women diagnosed with knee osteoarthritis. Postmenopause is defined as the absence of menstruation for at least 12 consecutive months. Participants will be randomly assigned to either the study or control group using a computer-generated randomization sequence. Allocation concealment will be ensured using sealed opaque envelopes. Both participants and outcome assessors will be blinded to the treatment allocation. The physical therapist applying iontophoresis will not be involved in outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* • Postmenopausal women aged 50-70 years.

  * Clinical and radiographic diagnosis of knee osteoarthritis according to the American College of Rheumatology criteria.
  * Radiographic severity classified as Kellgren-Lawrence grade II or III.
  * Chronic knee pain for a duration of at least 3 months.
  * Pain intensity ≥4 on the Visual Analog Scale.
  * Ability to ambulate independently with or without assistive devices.
  * Ability to understand and follow instructions.
  * Willingness to participate and provide written informed consent.

Exclusion Criteria:

* • Severe knee osteoarthritis (Kellgren-Lawrence grade IV).

  * History of knee surgery or intra-articular injections within the previous 6 months.
  * Presence of inflammatory rheumatic diseases such as rheumatoid arthritis or gout.
  * Neurological disorders affecting lower limb function.
  * Uncontrolled metabolic, cardiovascular, or systemic diseases.
  * Current or recent use of metformin or other antidiabetic medications.
  * Skin lesions, infections, or hypersensitivity at the iontophoresis site.
  * Contraindications to electrotherapy such as pacemakers or implanted electronic devices.
  * Body mass index ≥35 kg/m².
  * Participation in another clinical trial within the last 3 months.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal Women
Enrollment: 68 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | at baseline, after 6 weeks and after 12 weeks
  assessed using the Visual Analog Scale.
Functional status | at baseline, after 6 weeks and after 12 weeks
  assessed using the WOMAC index

CONTACTS AND LOCATIONS:
Locations (1):
- Badr University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Bannuru RR, Osani MC, Vaysbrot EE, et al. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis and Cartilage. 2019;27(11):1578-1589. 2. Kolasinski SL, Neogi T, Hochberg MC, et al. 2020 American College of Rheumatology guideline for the management of osteoarthritis of the hand, hip, and knee. Arthritis Care & Research. 2020;72(2):149-162. 3. Quicke JG, Foster NE, Ogollah RO, et al. Supervised exercise therapy for knee osteoarthritis: A randomized controlled trial. Ann Rheum Dis. 2022;81(3):336-343. 4. Wang Y, Hussain SM, Wluka AE, et al. Effect of exercise therapy on knee osteoarthritis: Systematic review and meta-analysis. Arthritis Res Ther. 2021;23:147. 5. Zhang W, Doherty M, Peat G, et al. EULAR evidence-based recommendations for knee osteoarthritis management. Ann Rheum Dis. 2020;79(6):685-699.